CLINICAL TRIAL: NCT03495544
Title: Comparative, Multicenter Study Estimating Association Between Germline DNA-repair Genes Mutations and PD-L1 Expression Level in Breast Cancer
Brief Title: Study Estimating Association Between Germline Mutations and PD-L1 Expression in Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tatarstan Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: ESR-17-12934
Record Dates: First submitted 2018-03-15; First posted 2018-04-12 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Hereditary Breast Cancer
MeSH Terms: conditions — Breast Cancer, Familial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hereditary BC: Pathogenic germline mutations in DNA-repair genes (TP53 MLH1 MSH2 MSH6 PMS2 EPCAM APC MUTYH CDKN2A CDK4 ATM KIT PDGFRA CDH1 CTNNA1 PRSS1 SPINK1 BRCA1 BRCA2 FANCI FANCL PALB2 RAD51B RAD51C RAD54L RAD51D CHEK1 CHEK2 CDK12 BRIP1 PPP2R2A BARD1 PARP1 STK11 XRCC3)
  Interventions: Diagnostic Test: PD-L1 expression
- Sporadic BC: Without germline mutations in DNA-repair genes (TP53 MLH1 MSH2 MSH6 PMS2 EPCAM APC MUTYH CDKN2A CDK4 ATM KIT PDGFRA CDH1 CTNNA1 PRSS1 SPINK1 BRCA1 BRCA2 FANCI FANCL PALB2 RAD51B RAD51C RAD54L RAD51D CHEK1 CHEK2 CDK12 BRIP1 PPP2R2A BARD1 PARP1 STK11 XRCC3)
  Interventions: Diagnostic Test: PD-L1 expression

INTERVENTIONS:
Diagnostic Test: PD-L1 expression — IHC testing of PD-L1 expression level in tumor tissue samples

SUMMARY:
This is a multicentre, non-interventional, prospective study to be carried out in representative oncology departments / institutions in order to determine the association between the presence of germline DNA-repair genes mutations and PD-L1 expression level in tumour and immune cells in breast cancer. No additional procedures besides those already used in the routine clinical practice will be applied to the patients.

DETAILED DESCRIPTION:
Breast cancer (BC) occupies the first place among malignancy in females (29.9% of all tumors in female patients in Russian Federation in 2015) [1].

One of the most perspective direction of the oncotherapy is anticancer immunotherapy - employment of inhibitors of immune checkpoints. Immune checkpoints inhibitors (such as anti-PD-1 and anti-PD-L1 antibodies) have shown good clinical efficiency in clinical research to cure such malignant tumor with high mutation load, as melanoma, lung cancer, and others.

One of the hypothesis of such effect states that, usually, more cancer neoantigens are synthetized in the tumors with high mutation load (driven by genome instability), causing severe lymphoid infiltration [2-3]. This situation is balanced by overexpression of such inhibitors of the immune response as PD-1 and PD-L1 [4 - 6].

Breast cancer - is relatively heterogenic tumor, with different genetic, morphological and phenotypic forms.

Despite relatively low expression of PD-L1 in BC in general, there are reasons to believe that genetic instability, driven by mutations in genes involved in DNA repair, can increase the immunogenicity and, thus, the expression of PD-L1 in BC.

To date, it is widely accepted that 5-10% of BC cases are represented by hereditary types, i.e. mediated by germline pathogenic mutations in genes of DNA reparation pathways. Hereditary breast cancer (HBC), as well as ovarian cancer (OC), сaused by mutations in genes BRCA1, BRCA2, CHEK2, TP53 и PTEN, and others. Thus, one of the promising directions here is to understand the inter-relation among germline pathogenic mutations associated with HBC, and activity of PD-L1. It would allow to optimize selection of anti-PD-L1 therapy, by forming group of patients (matching criteria of HBC) with high level of PD-L1 expression in cancer cells and tumor-infiltrating lymphocytes.

ELIGIBILITY:
Inclusion Criteria:

* 1. The voluntary obtained informed consent signed by both the subject and the investigator.

  2. Females 18 years age or more. 3. Histologically confirmed BC with known hormone receptors and HER2neu receptors status, Grade of tumor, diagnosed before enrolment into the study.

  4. Availability of FFPE tissue samples received prior to any type of antitumor treatment start. Tumour tissue samples must be satisfied IHC requirements for PD-L1 testing.

  5. Ability of blood samples receiving for NGS germline mutations testing. 6. Completed medical records (stage, receptors status, demographic data)

Exclusion Criteria:

* Any evidence of uncontrolled system pathology, active infections, active bleeding diathesis, renal graft, including virus hepatitis B, C or HIV.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients, female aged between 18-80yrs with breast cancer
Sampling Method: Probability Sample
Enrollment: 390 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-03-17 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of PD-L1 expression in breast cancer | January 2018-January 2019
  Number of samples of PD-L1 high expression in tumor and immune cells in FFPE breast tumor tissue and number of samples of PD-L1 low expression in tumor and immune cells in FFPE breast tumor tissue .
  The report will be represented as "PD-L1 high" or "PD-L1 low".

SECONDARY OUTCOMES:
Diagnostic performance of inherited gene mutations in breast cancer | January 2018-January 2019
  Mutations will be determined by "pathogenic" and "non pathogenic". Number of samples with "pathogenic" and "non pathogenic" mutations .
Association between germline DNA-repair genes mutations and PD-L1 expression level in in breast cancer | January 2018-January 2019
  To reveal the differences (percentages) of PD-L1 high tumor rate between patients with hereditary BC ( pathogenic mutations) who have clinically significant germline mutations in DNA-repair genes (HR- deficiency) and patients with sporadic BC without such mutations (non pathogenic mutations).

CONTACTS AND LOCATIONS:
Locations (1):
- Tatarstan Cancer Cente, Kazan', Tatarstan Republic, Russia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT03495544/Prot_SAP_000.pdf
  • Informed Consent Form (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT03495544/ICF_001.pdf